CLINICAL TRIAL: NCT01522209
Title: Value of Contrast Enhanced Intraoperative Ultrasound Compared to Preoperative CEUS, CT and MRT in the Treatment of Colorectal Liver Metastases.
Brief Title: Detection Rate of Liver Metastases With Contrast Enhanced Intraoperative Ultrasound Compared to Regular Imaging
Acronym: CEIOUS-Liver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asklepios Kliniken Hamburg GmbH (Other)
Responsible Party: Principal Investigator, Dr. Gregor A. Stavrou, Principal Investigator, Asklepios Kliniken Hamburg GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Asklepios
Record Dates: First submitted 2012-01-03; First posted 2012-01-31 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Colon Cancer Liver Metastasis; Contrast Enhances Intraoperative Ultrasound; Imaging for Liver Cancer; Imaging for Liver Metastasis
Keywords: CRLM; Primovist MRI; CEIOUS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Liver Surgery — R0 Resection of Liver Metastases after Planning with preoperative imaging data and comparison with intraoperative contrast enhanced ultrasound
Device: Contrast Enhanced Ultrasound — The contrast enhanced Ultrasound imaging is performed before and during the operation using Sonovue contrast agent (2.5ml iv preop, 4.5ml iv intraop)
Radiation: CT Scan (standard) — A staging CT of the liver/abdomen with the minimal possible dosage for aquiring sufficent triphasic data in a 64-line helical scan
Radiation: Primovist MRI (3 Tesla) — an MRI scan of the liver with Primovist contrast agent including late phase as addition to the preop staging according to the protocol

SUMMARY:
The study compares the established imaging techniques (CT, MRT, Contrast Ultrasound) with the new method of intraoperative contrast enhanced ultrasound to compare all methods for their rate of detection of colorectal liver metastasis.

DETAILED DESCRIPTION:
1. Introduction: The surgical resection of colorectal liver metastases is the only curative therapy for those patients (1). Because a major part of those patients become diagnosed in a technical irresectable stadium, most patients primary get a chemotherapy to reach a secondary resection (2). Especially for this group of patients an effective preoperative staging is necessary to know the exact number and location of the liver metastases. Standard imaging is abdominal CT with a contrast medium, lately it is also possible to create a 3D analysis based on vasculatory territories out of the 2D data (3) (4). Alternatively MRI imaging can be used as well, but because of its defiency in the imaging of vascular anatomy it is only partly suited for the surgical planning and resection. By now the contrast enhanced sonography has been further developed and can be used for dignity evaluation of leasions. Depending on the examiner it can provide very useful informations (5). Because of the intraoperative ultrasound is the most sensitive and specific diagnosic procedure (6), the intraoperative use of contrast medium ultrasound seems to suggest itself. As the necessary ultrasonic probes weren't avaiable until now, only a few experiences have been made yet (7).

Aim of the study is to compare the value of all described methods considering the detection rate of colorectal metastases, including the by now available intraoperative cm-ultrasound. From the comparison of all modern methods (64-line doublehelix CT, 3D virtual operation planning, 3 tesla Primovist-MRI, pre- and intraoperative contrast enhanced sonography) we aim to get a reliable recommendation for the preoperative necessary staging.

1. Background: state of research/ scientific arguementation/ leading question In the last 20 years, the surgery of colorectal liver metastases has developed a lot (8,9,10,11). In centers even complex surgeries can be done with a mortality of 0,1% and with a morbidity of 15%. Today, neither the number, nor the localisation of metastases or an extrahepatic tumour growth is decisive for a resection, but the fact, if there is a possibilty for a complete tumor excision (12). Especially because of the further developement of neoadjuvant (13) and adjuvant (14) chemotherapeutics on the one hand and the technical developement (portal embolisation (15), two-time resection (16), virtual operation planning (4), navigated surgery (17)) on the other hand enlarged the number of patients becoming resectable secondarily.

The demand on preoperative imaging increased with the technical and therapeutical developements. In surgical and technical prospect the abdomen CT imaging is still standard in surgery planning, because besides the tumor imaging, the good vascular anatomy imaging enables a surgical strategy (5). Today, 2D CT data can be used to create a 3D imaging of the liver and its vascularisation to plan a virtual surgery beneffiting especially the most complex surgeries (18). Because of the distinct better resolution of a lesion, MRI imaging of the liver has a high significance in literature and allows radiologists a higher quality of their diagnosis (19), but does not obligatory ease the surgery planning for the surgeon (20). A comparing study in a surgeons point of view could show a equal validity of both modalities (21). Interestingly, the mentionend studies showed that the detection of metastases in altered liver tissue (fatty degeneration/ status post chemotherapy) is reduced. In these difficult cases the CE-sonography gives the decisive informations (22). The practical disadvantage is the dependence on the examiner.

Intraoperative sonography is the gold standard procedure during the operation, additional leasions can be detected which may change the resection strategy (6). Even if there are only a few experiences with intraoperative ultrasonic probes that are able to do contrast enhancment, we assume an advantage of the use of contrast medium sonography (23) in the operation room. The yet published data is not enough for a ensured evidence.

In our point of view it is necessary to carry out a prospective study comparing all available state of the art imaging methods and adding the intraoperative contrast enhanced ultrasound to validate it´s effect.

In times of limited resources it becomes more and more important with a lot of difference in the costs for the imaging modalities to define an optimal staging for these complex patients that at the same time has enough value for the surgeon to go forward with an operation.

3. Design The Study is concepted as a prospective, monocentric and controlled observational study.

4. Primary Endpoints: the detection of the liver metastases intraoperative and the comparison with the preoperative information. Secondary endpoints : comparison of the detection-rates of all the imaging methods, comparison of the sensitivity of all the imaging methods and comparison of the specificity of all imaging methods.

5. Caseload discussion and statistical Analysis: As the primary target figure the number of metastases detected during the operation using ultrasound and CT/MRI are taken into consideration.

It has to be shown that the average number of the liver metastases that have been detected using the two procedures CE-IOUS and CT/MRI are different. On average using the CE-IOUS method for the patient sample detects 1.95 metastases, the pre surgery detects 1.54 metastases using CT/MRI.

The standard deviation between the detected metastasis is 1.10.

The null- and alternative hypothesis of the key question is:

H0: the two procedures CE-IOUS and CT/MRI detect the same number of metastases, H1: CE-IOUS and CT/MRI detect unequal numbers of metastases. It has been presumed that the CE-IOUS method is more successful in detection of the metastases . To test the two-sided question a paired T-test with an average difference of 0 regarding the absolute detection-number on a significance level of 5% with a stastistical power of 90% will be used.

To be able to prove the difference between the two methods a number of 78 patients must be evaluated. With respect to the 20% rate of drop-outs 98 patients were recruited.

6. Patient population: 98 patient are supposed to be included in this study. Operation and execution: in the first contact we will explain to our patients the research plan. The case will be discussed at our interdisciplinary tumor conference. The next step is imaging with CT abdomen and contrast medium sonography. Data of the CT will be finished of for a 3D surgery planning.

In the next step we carry out a MRI of the liver. Preoperative all imaging methods will be compared. Thus we plan an operative strategy. Intraoperative the regular sonography will be supplemented by contrast media (this leads to an extention of the 4 hour surgery by 10 minutes. Afterwards we carry out the liver resection.

Data of all the imaging techniques with regard to detection of metastases, species delineation of the leasion, preoperative resection strategies as well as intraoperative changes of the resection strategies will be collected in a data base. Patients will be provided with care immediately after they are discharged. Therefore, every six months they will be send to our special consultation. The data we gain will subsequently be tested for statistical significance and will then be evaluated (MS Excel, SPSS). The results will be published in medical literature.

For the trail, we plan to use the data of patients in a period of 18 months. Our hospital carries out about 80 liver resections every year hence we should be able to collect 98 patients with colorectal metastases. With this amount we can gain a meaningful analysis.

7. There are risks and additional strain for patients by the additional administration of contrast media during MRI imaging. There is a possibility that it leads to severe reaction of the body (<1:100.000) which can be treated medicinal.

In our opinion, there is no risk due to the elongation of the about 4 hour enduring surgery for 10 minutes because of the contrast media sonography. This is because of the surgical morbidity by liver resection not because of the procedure of the sonography.

8. Possible benefit for the patient: With the possibility of having an optimal staging sequence with high reliability using todays imaging methods not only can more and more patients benefit from therapeutic measures with high chances of cure but many might also be spared from unnecessary surgeries.

In medical literature there is still a controversary discussion about the ideal imaging modality in liver surgery. Here, different angles of view encounter the same problem (surgical/radiological view) both availability of methods (CT/MRI) and their costs. For the advancement of the always more complex and interdisciplinary stamped treatment strategies of colorectal liver metastases it is vital to use a reliable imaging method and respectively for a high significance a combination of methods. The intraoperative contrast media sonography promises a significant benefit in the detection of leasions which have not been detected so far. In the future patients may benefit a lot from it and thus get a better prognosis. The up to now existing data are not sufficient. Therefore, from our point of view, it is very important to consider the comparative consideration of all modalities.

9. Abruption criteria revocation of accordance of attendance of a trail through the patient and factors, which do not allow a surgical intervention.

10. Voluntary attendance and countermand of the accordance The patient's attendance on this project is voluntary. The decision of taking part or not, does not interfere with the right to sanitary protection or other attainments. The decision of taking part or not does not intervene with the Health protection claim or other services to which the patients are entitled. The patients in no way denounce their legal claims or rights by taking part in this study. When the patients make a decision to take part they are granted the power to withdraw or revoke their consent and abort their participation.

11. Ethical basis of this study is carried out according to the declaration of the 18th world medical association of Helsinki, Finland 1964 and the later revisions. The study will be presented to the Ethic committee of Hamburg for careerlegal counceling. Possible subsequent changes will be presented to the Ethic committee for assessment.

12. Data privacy that have been collected according to the patients consent, particularly results, underlie discretion and the data privacy assignation. They will be recorded and saved in paper format and data medium in the Asklepios clinic Barmbek, department of general and visceral surgery. The use of these Data is carried out pseudonymously. A transmission of the data for research purposes will also be done pseudonymously. The same rule applies to publication of the study- and scientific results.

These patients have the right to demand information regarding their personal data and possible personal results. Where appropriate the head of the study or the scientific manager will make the decision.

(The recording and saving of the data will take place for a period of ten years.) In case of revocation of the consent the already collected data will be further used in this format.

The Literature is found under Citations

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Age > 18 years All Patients presenting with Colorectal Liver Metastasis indicated for Liver Surgery in the study period

Exclusion Criteria:

* No Informed Consent Possible Pregnancy Patients with hereditary diseases of the metabolic system Liver Cirrhosis CHILD B and C Renal Insufficiency defined as Kreatinin >2,5 mg/dl PAtients enrolled in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Detection of Liver Metastasis during Operation | During Operation
  Intraoperative Rate of Detection of Liver Metastasis compared to preoperative Imaging Analysis

SECONDARY OUTCOMES:
Comparison of Detection Rate for Liver Metastases of all imaging modalities | 1 Week after Operation
Comparison of Sensitivity of all imaging modalities | one Year
Comparison of Specicivity of all imaging modalities | one year

CONTACTS AND LOCATIONS:
Overall Officials: Gregor A Stavrou, Dr.med, Principal Investigator — Dpt. of General and Visceral Surgery, Asklepios Hospital Barmbek, Hamburg, Germany
Locations (1):
- Asklepios Hospital Barmbek, Hamburg, Hamburg, Germany

REFERENCES:
- [Background] Lupinacci R, Penna C, Nordlinger B. Hepatectomy for resectable colorectal cancer metastases--indicators of prognosis, definition of resectability, techniques and outcomes. Surg Oncol Clin N Am. 2007 Jul;16(3):493-506, vii-viii. doi: 10.1016/j.soc.2007.04.014. PMID 17606190
- [Background] Nordlinger B, Van Cutsem E, Rougier P, Kohne CH, Ychou M, Sobrero A, Adam R, Arvidsson D, Carrato A, Georgoulias V, Giuliante F, Glimelius B, Golling M, Gruenberger T, Tabernero J, Wasan H, Poston G; European Colorectal Metastases Treatment Group. Does chemotherapy prior to liver resection increase the potential for cure in patients with metastatic colorectal cancer? A report from the European Colorectal Metastases Treatment Group. Eur J Cancer. 2007 Sep;43(14):2037-45. doi: 10.1016/j.ejca.2007.07.017. Epub 2007 Sep 4. PMID 17766104
- [Background] Oldhafer KJ, Hogemann D, Stamm G, Raab R, Peitgen HO, Galanski M. [3-dimensional (3-D) visualization of the liver for planning extensive liver resections]. Chirurg. 1999 Mar;70(3):233-8. doi: 10.1007/s001040050636. German. PMID 10230533
- [Background] Lang H, Radtke A, Hindennach M, Schroeder T, Fruhauf NR, Malago M, Bourquain H, Peitgen HO, Oldhafer KJ, Broelsch CE. Impact of virtual tumor resection and computer-assisted risk analysis on operation planning and intraoperative strategy in major hepatic resection. Arch Surg. 2005 Jul;140(7):629-38; discussion 638. doi: 10.1001/archsurg.140.7.629. PMID 16027326
- [Background] Ong KO, Leen E. Radiological staging of colorectal liver metastases. Surg Oncol. 2007 Jul;16(1):7-14. doi: 10.1016/j.suronc.2007.04.001. Epub 2007 May 11. PMID 17499498
- [Background] Cervone A, Sardi A, Conaway GL. Intraoperative ultrasound (IOUS) is essential in the management of metastatic colorectal liver lesions. Am Surg. 2000 Jul;66(7):611-5. PMID 10917467
- [Background] Nakano H, Ishida Y, Hatakeyama T, Sakuraba K, Hayashi M, Sakurai O, Hataya K. Contrast-enhanced intraoperative ultrasonography equipped with late Kupffer-phase image obtained by sonazoid in patients with colorectal liver metastases. World J Gastroenterol. 2008 May 28;14(20):3207-11. doi: 10.3748/wjg.14.3207. PMID 18506927
- [Background] Scheele J, Stangl R, Altendorf-Hofmann A. Hepatic metastases from colorectal carcinoma: impact of surgical resection on the natural history. Br J Surg. 1990 Nov;77(11):1241-6. doi: 10.1002/bjs.1800771115. PMID 2253003
- [Background] Scheele J, Stang R, Altendorf-Hofmann A, Paul M. Resection of colorectal liver metastases. World J Surg. 1995 Jan-Feb;19(1):59-71. doi: 10.1007/BF00316981. PMID 7740812
- [Background] Belghiti J, Hiramatsu K, Benoist S, Massault P, Sauvanet A, Farges O. Seven hundred forty-seven hepatectomies in the 1990s: an update to evaluate the actual risk of liver resection. J Am Coll Surg. 2000 Jul;191(1):38-46. doi: 10.1016/s1072-7515(00)00261-1. PMID 10898182
- [Background] Benoist S, Nordlinger B. Neoadjuvant treatment before resection of liver metastases. Eur J Surg Oncol. 2007 Dec;33 Suppl 2:S35-41. doi: 10.1016/j.ejso.2007.09.022. Epub 2007 Nov 5. PMID 17981428
- [Background] Pawlik TM, Schulick RD, Choti MA. Expanding criteria for resectability of colorectal liver metastases. Oncologist. 2008 Jan;13(1):51-64. doi: 10.1634/theoncologist.2007-0142. PMID 18245012
- [Background] Folprecht G, Gruenberger T, Bechstein WO, Raab HR, Lordick F, Hartmann JT, Lang H, Frilling A, Stoehlmacher J, Weitz J, Konopke R, Stroszczynski C, Liersch T, Ockert D, Herrmann T, Goekkurt E, Parisi F, Kohne CH. Tumour response and secondary resectability of colorectal liver metastases following neoadjuvant chemotherapy with cetuximab: the CELIM randomised phase 2 trial. Lancet Oncol. 2010 Jan;11(1):38-47. doi: 10.1016/S1470-2045(09)70330-4. Epub 2009 Nov 26. PMID 19942479
- [Background] Portier G, Elias D, Bouche O, Rougier P, Bosset JF, Saric J, Belghiti J, Piedbois P, Guimbaud R, Nordlinger B, Bugat R, Lazorthes F, Bedenne L. Multicenter randomized trial of adjuvant fluorouracil and folinic acid compared with surgery alone after resection of colorectal liver metastases: FFCD ACHBTH AURC 9002 trial. J Clin Oncol. 2006 Nov 1;24(31):4976-82. doi: 10.1200/JCO.2006.06.8353. PMID 17075115
- [Background] Abdalla EK, Hicks ME, Vauthey JN. Portal vein embolization: rationale, technique and future prospects. Br J Surg. 2001 Feb;88(2):165-75. doi: 10.1046/j.1365-2168.2001.01658.x. PMID 11167863
- [Background] Wicherts DA, Miller R, de Haas RJ, Bitsakou G, Vibert E, Veilhan LA, Azoulay D, Bismuth H, Castaing D, Adam R. Long-term results of two-stage hepatectomy for irresectable colorectal cancer liver metastases. Ann Surg. 2008 Dec;248(6):994-1005. doi: 10.1097/SLA.0b013e3181907fd9. PMID 19092344
- [Background] Oldhafer KJ, Stavrou GA, Prause G, Peitgen HO, Lueth TC, Weber S. How to operate a liver tumor you cannot see. Langenbecks Arch Surg. 2009 May;394(3):489-94. doi: 10.1007/s00423-009-0469-9. Epub 2009 Mar 12. PMID 19280221
- [Background] Preim B, Bourquain H, Selle D, Oldhafer KJ. Resection Proposals for Oncologic Liver Surgery based on Vascular Territories. 2002 Mar. 8;
- [Background] Robinson P. The early detection of liver metastases. Cancer Imaging. 2002;
- [Background] Gaa J, Wieder H, Schwaiger M, Rummeny EJ. [Modern imaging for liver metastases from colorectal tumors]. Chirurg. 2005 Jun;76(6):525-6, 528-34. doi: 10.1007/s00104-005-1031-0. German. PMID 15875145
- [Background] Bhattacharjya S, Bhattacharjya T, Baber S, Tibballs JM, Watkinson AF, Davidson BR. Prospective study of contrast-enhanced computed tomography, computed tomography during arterioportography, and magnetic resonance imaging for staging colorectal liver metastases for liver resection. Br J Surg. 2004 Oct;91(10):1361-9. doi: 10.1002/bjs.4699. PMID 15376205
- [Background] Konopke R, Kersting S, Bergert H, Bloomenthal A, Gastmeier J, Saeger HD, Bunk A. Contrast-enhanced ultrasonography to detect liver metastases : a prospective trial to compare transcutaneous unenhanced and contrast-enhanced ultrasonography in patients undergoing laparotomy. Int J Colorectal Dis. 2007 Feb;22(2):201-7. doi: 10.1007/s00384-006-0134-5. Epub 2006 May 30. PMID 16733650
- [Background] Shah AJ, Callaway M, Thomas MG, Finch-Jones MD. Contrast-enhanced intraoperative ultrasound improves detection of liver metastases during surgery for primary colorectal cancer. HPB (Oxford). 2010 Apr;12(3):181-7. doi: 10.1111/j.1477-2574.2009.00141.x. PMID 20590885
- [Derived] Stavrou GA, Stang A, Raptis DA, Schadde E, Zeile M, Bruning R, Wagner KC, Huber TM, Oldhafer KJ. Intraoperative (Contrast-Enhanced) Ultrasound Has the Highest Diagnostic Accuracy of Any Imaging Modality in Resection of Colorectal Liver Metastases. J Gastrointest Surg. 2021 Dec;25(12):3160-3169. doi: 10.1007/s11605-021-04925-2. Epub 2021 Jun 22. PMID 34159555